CLINICAL TRIAL: NCT06005233
Title: Smartwatches for Detection of Atrial Fibrillation (AFib) in Secondary Prevention of Cryptogenic Stroke - WATCH AFib A Prospective, Intraindividual-controlled, Multicenter Clinical Study
Brief Title: Smartwatches for Detection of Atrial Fibrillation (AFib) in Secondary Prevention of Cryptogenic Stroke
Acronym: WATCH AFib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20230726
Record Dates: First submitted 2023-08-01; First posted 2023-08-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke, Cryptogenic; Transient Ischemic Attack; Atrial Fibrillation
Keywords: Smartwatch; Ischemic stroke; atrial fibrillation
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective, intraindividual-controlled, multicenter clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of Smartwatch (Experimental): Application of smartwatch in addition to an implanted event recorder. Follow-up of 6 months
  Interventions: Device: Smartwatch

INTERVENTIONS:
Device: Smartwatch — Smartwatch with PPG- and 1-lead ECG derived analysis of cardiac arrhythmia. Analysis will be performed centrally at the Cardiology Core Lab at the Klinikum Rechts der Isar.

SUMMARY:
Scientific Background: In secondary prevention of ischemic stroke, detection of atrial fibrillation (AFib) and subsequent anticoagulation therapy reduce the risk of recurrent stroke by approximately 60%. Prolonged electrocardiogram (ECG) monitoring up to 6 months significantly increases detection of AFib in cryptogenic stroke. Wearables like smartwatches have recently been shown to adequately detect AFib in the general population. Thus, prolonged ECG monitoring after cryptogenic ischemic stroke or transient ischemic attack (TIA) using a smartwatch could lead to a reduction of recurrent stroke by prompting adequate anticoagulation therapy and may constitute a cost-effective, non-invasive, and broadly-available alternative to the current standard of care.

Hypothesis: The investigators hypothesize that AFib detection via smartwatch in patients with cryptogenic TIA or ischemic stroke is accurate compared to an implantable event recorder.

Methods: The investigators introduce a prospective, intraindividual-controlled, multicentre clinical study in patients with cryptogenic ischemic stroke or TIA. In addition to an implanted event recorder as indicated by clinical standard, included patients receive a smartwatch for detection of AFib. ECG-data from smartwatches will be continuously monitored by two independent cardiologists. As soon as AFib is confirmed, a doctoral appointment is set to evaluate start of anticoagulation. The follow-up period will be six months. The study consists of four study visits: a baseline visit, two phone visits at one and three months, and an end of trial visit at six months.

Primary Objective: To compare smartwatch and event recorder based analysis for sensitivity and specificity of AFib detection per patient after six months

DETAILED DESCRIPTION:
Ischemic stroke is worldwide the second most frequent cause of death and disability and has a lifetime risk of approximately 25%. In the secondary prevention of ischemic stroke, detection of atrial fibrillation (AFib) and subsequent anticoagulation therapy reduce the risk of recurrent stroke by approximately 60%. Cryptogenic stroke is defined as ischemic stroke for which no probable cause is found despite a full standard evaluation and comprises 25% of all ischemic strokes. Prolonged electrocardiogram (ECG) monitoring for 30 days to 6 months significantly increases the detection of occult paroxysmal AFib in cryptogenic stroke, which is present in 9 - 16%. Thus, prolonged ECG monitoring is likely to lead to a reduction of recurrent stroke by prompting adequate anticoagulation therapy.

Still, prolonged AFib screening after stroke is currently suboptimal due to a limitation of resources, loss to follow-up, invasiveness of procedures, and costs. Wearables like smartwatches have recently been shown to adequately detect AFib in the general population. Sensitivity and specificity of AFib detection compared to ECG-based diagnosis is high (93-98% and 90-98%, respectively). Compared to implantable Event Recorders, smartwatch based AFib diagnosis in the general population exhibits a sensitivity of 97.5% for AFib episodes >1h and a sensitivity of 100% for AFib detection per patient.

The investigators hypothesize that AFib detection via smartwatch in patients suffering from cryptogenic transient ischemic attack (TIA) or ischemic stroke is accurate for AFib detection compared to an implantable Event Recorder and might therefore be a non-invasive, cost-effective, widely available alternative, which could potentially change the current standard of post-stroke care.

The primary objective is to assess whether AFib detection via smartwatch in patients suffering from cryptogenic TIA/ ischemic stroke is accurate in comparison to implantable Event Recorders. This will be assessed by sensitivity and specificity of AFib detection per patient after six months. The investigators aim on a comparison of smartwatch based, continuous, automated, cardiologist supervised rhythm analysis of photoplethysmography (PPG)- signal and patient activated 1-lead ECG with Event Recorder based, continuous, automated ECG rhythm analysis.

This is a prospective, intraindividual-controlled, multicenter clinical study.

The study population includes patients with cryptogenic TIA or ischemic stroke and known risk factors for the presence of paroxysmal AFib (see inclusion criteria; CHA2DS2VASc score ≥4, Atrial runs, Left atrial size > 45mm, Left atrial appendage flow ≤ 0.2m/s).

In addition to an implanted Event Recorder according to clinical standard, patients receive a smartwatch. Smartwatch- and Event Recorder-derived heart rhythm are daily uploaded and ana-lyzed by the cardiologists at the Cardiology Core Lab at the Department of Internal Medicine I, Klinikum rechts der Isar, Munich. The obtained data on cardiac arrhythmia will be assessable for each study site in consultation with the Cardiology Core Lab. In case of an arrhythmic event, the obtained data on duration, source of information (e.g., smartwatch PPG signal, smartwatch 1-lead ECG, Event Recorder) will be implemented in the eCRF by the Cardiology Core Lab.

In parallel, the study consists of a total of four visits. The baseline visit (Visit 0) may take place within the clinical setting of the acute stroke work up. A table containing a detailed plan of the data to be collected will be provided. Furtherly, the implementation and set-up of the smart-watch will take place within the baseline visit. A manual will be provided for each study center and patient to correctly set up and instruct on the usage of the smartwatch. The second and third visit (Visit 1, Visit 2) constitute phone-visits at one and three months with a tolerated time deviation of one week. The last visit at the end of the study (Visit 3) will be performed at six months with a tolerated time deviation of three weeks. This visit will take place at each pa-tient's study center. A table containing a detailed plan of the data to be collected will be pro-vided for each study center.

The first patient is planned to be included approximately in the third quarter of 2023 and the last patient approximately in the first quarter of 2025. Accordingly, the last patient will exit the study ('last patient last visit') approximately by the end of 2025.

The clinical study will be carried out in accordance with the study protocol and the principles of the Declaration of Helsinki by the World Medical Association and specific applicable national ethical and regulatory requirements.

All patients included in the clinical study will receive standard of care for cryptogenic TIA/ is-chemic stroke. The clinical study protocol does not interfere with generally accepted standards in post stroke care and local SOPs .The applied smartwatch is CE-certified as a medical device for AFib detection. As the study intervention consists in simply wearing a smartwatch (and phone visits are implemented at one and three months), we expect no safety risk for study partici-pants.

ELIGIBILITY:
Inclusion Criteria:

* Implanted Event Recorder with telemedicinal function (e.g., Biotronik BioMon 3m ProMRI HomeMon or similar)
* Cryptogenic stroke (within the last six month) after full standard evaluation:

  * Stroke detected by computed tomography (CT) or magnetic resonance imaging (MRI) that is not lacunar (lacunar is defined as a subcortical infarct in the distribution of the small, penetrating cerebral arteries whose largest dimension is ≤1.5 cm on CT or ≤2.0 cm on MRI diffusion images)
  * Absence of extracranial or intracranial atherosclerosis causing ≥50 percent luminal stenosis of the artery supplying the area of ischemia
  * No major-risk cardioembolic source of embolism (i.e., no permanent or paroxysmal atrial fibrillation, sustained atrial flutter, intracardiac thrombus, prosthetic cardiac valve, atrial myxoma or other cardiac tumors, high-grade mitral valve stenosis, recent (within four weeks) myocardial infarction, left ventricular ejection fraction <30 percent, valvular vegetations, or infective endocarditis)
  * No other specific cause of stroke identified (e.g., arteritis, dissection, migraine, vasospasm, drug abuse)
  * No paroxysmal atrial fibrillation in 72h of in-hospital ECG-monitoring, including at least one Holter- ECG for 24 hours.
* Cryptogenic TIA with definite cortical syndrome (aphasia, neglect or homonymous hemianopia) (within the last six month) after full standard evaluation (see above)
* Age: ≥40 yrs.
* At least one of the following risk factors:

  * CHA2DS2VASc score ≥4
  * Atrial runs
  * Left atrial size > 45mm
  * Left atrial appendage flow ≤ 0.2m/s
* No contraindication for anticoagulant therapy after acute phase of stroke
* Written informed consent by patient or authorized caregiver

Exclusion Criteria:

* Patient is not able to perform 1-lead ECG recording with smartwatch
* Patient possesses no smartphone (iOS version ≥10.0 or Android)
* Implanted pacemaker or cardioverter defibrillator (ICD)
* Pregnancy and breastfeeding period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of AFib Detection | From baseline visit (V0) to the last follow-up at visit (V3) at six months
  To estimate and compare sensitivity and specificity for AFib detection per patient after six months (Comparison of smartwatch based, continuous, automated, cardiologist supervised rhythm analysis of photoplethysmography (PPG)- signal and patient activated 1-lead ECG with Event Recorder based, continuous, automated ECG rhythm analysis).

SECONDARY OUTCOMES:
To estimate and compare the positive and negative predictive values for AFib detection per patient | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Sensitivity and specificity for AFib detection of the automated PPG-signal rhythm analysis | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Sensitivity and specificity for the detection of any AFib episode | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Sensitivity for the detection of AFib episodes >1 hour | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Sensitivity and specificity of AFib detection per recorded/ per analyzable time (i.e., intervals in which the watch is actually worn/records an analyzable signal; per-protocol analysis) | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Specificity for episodes of sinus rhythms >1 hour | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Stroke and TIA recurrence within six months | From baseline visit (V0) to the last follow-up at visit (V3) at six months
  Stroke or TIA recurrence in the clinical follop-up visits at 1, 3 and 6 months
Subgroup analysis: accuracy in severely affected patients (i.e., National Institute of Health Stroke Scale (NIHSS) ≥8) | From baseline visit (V0) to the last follow-up at visit (V3) at six months
  NIHSS: 0-42 points, a higher score refers to the presence of more stroke related symtpoms/ worse outcome
Exploratory endpoint: Acceptance and practicability of smartwatches for AFib detection | From baseline visit (V0) to the last follow-up at visit (V3) at six months
  self-designed questionnaire
Exploratory endpoint: AFib burden/ patient | From baseline visit (V0) to the last follow-up at visit (V3) at six months
  Duration of AFib episodes/ Duration of Sinus rhythm
Exploratory endpoint: relevance of AFib risk factors | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Exploratory endpoint: AFib detection rates after one month and after six months and time to confirmed AFib diagnosis | From baseline visit (V0) to the last follow-up at visit (V3) at six months
Exploratory endpoint: count of AFib diagnoses | From baseline visit (V0) to the last follow-up at visit (V3) at six months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Technische Universität München, Munich, Germany

REFERENCES:
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Secondary prevention in non-rheumatic atrial fibrillation after transient ischaemic attack or minor stroke. EAFT (European Atrial Fibrillation Trial) Study Group. Lancet. 1993 Nov 20;342(8882):1255-62. PMID 7901582
- [Background] Hart RG, Pearce LA, Koudstaal PJ. Transient ischemic attacks in patients with atrial fibrillation: implications for secondary prevention: the European Atrial Fibrillation Trial and Stroke Prevention in Atrial Fibrillation III trial. Stroke. 2004 Apr;35(4):948-51. doi: 10.1161/01.STR.0000120741.34866.1D. Epub 2004 Feb 26. PMID 14988571
- [Background] Hart RG, Diener HC, Coutts SB, Easton JD, Granger CB, O'Donnell MJ, Sacco RL, Connolly SJ; Cryptogenic Stroke/ESUS International Working Group. Embolic strokes of undetermined source: the case for a new clinical construct. Lancet Neurol. 2014 Apr;13(4):429-38. doi: 10.1016/S1474-4422(13)70310-7. PMID 24646875
- [Background] Sanna T, Diener HC, Passman RS, Di Lazzaro V, Bernstein RA, Morillo CA, Rymer MM, Thijs V, Rogers T, Beckers F, Lindborg K, Brachmann J; CRYSTAL AF Investigators. Cryptogenic stroke and underlying atrial fibrillation. N Engl J Med. 2014 Jun 26;370(26):2478-86. doi: 10.1056/NEJMoa1313600. PMID 24963567
- [Background] Gladstone DJ, Spring M, Dorian P, Panzov V, Thorpe KE, Hall J, Vaid H, O'Donnell M, Laupacis A, Cote R, Sharma M, Blakely JA, Shuaib A, Hachinski V, Coutts SB, Sahlas DJ, Teal P, Yip S, Spence JD, Buck B, Verreault S, Casaubon LK, Penn A, Selchen D, Jin A, Howse D, Mehdiratta M, Boyle K, Aviv R, Kapral MK, Mamdani M; EMBRACE Investigators and Coordinators. Atrial fibrillation in patients with cryptogenic stroke. N Engl J Med. 2014 Jun 26;370(26):2467-77. doi: 10.1056/NEJMoa1311376. PMID 24963566
- [Background] Tsivgoulis G, Katsanos AH, Mac Grory B, Kohrmann M, Ricci BA, Tsioufis K, Cutting S, Krogias C, Schellinger PD, Campello AR, Cuadrado-Godia E, Gladstone DJ, Sanna T, Wachter R, Furie K, Alexandrov AV, Yaghi S. Prolonged Cardiac Rhythm Monitoring and Secondary Stroke Prevention in Patients With Cryptogenic Cerebral Ischemia. Stroke. 2019 Aug;50(8):2175-2180. doi: 10.1161/STROKEAHA.119.025169. Epub 2019 Jun 20. PMID 31216964
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Background] Tison GH, Sanchez JM, Ballinger B, Singh A, Olgin JE, Pletcher MJ, Vittinghoff E, Lee ES, Fan SM, Gladstone RA, Mikell C, Sohoni N, Hsieh J, Marcus GM. Passive Detection of Atrial Fibrillation Using a Commercially Available Smartwatch. JAMA Cardiol. 2018 May 1;3(5):409-416. doi: 10.1001/jamacardio.2018.0136. PMID 29562087
- [Background] Dorr M, Nohturfft V, Brasier N, Bosshard E, Djurdjevic A, Gross S, Raichle CJ, Rhinisperger M, Stockli R, Eckstein J. The WATCH AF Trial: SmartWATCHes for Detection of Atrial Fibrillation. JACC Clin Electrophysiol. 2019 Feb;5(2):199-208. doi: 10.1016/j.jacep.2018.10.006. Epub 2018 Nov 28. PMID 30784691
- [Background] Wasserlauf J, You C, Patel R, Valys A, Albert D, Passman R. Smartwatch Performance for the Detection and Quantification of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2019 Jun;12(6):e006834. doi: 10.1161/CIRCEP.118.006834. PMID 31113234
- [Background] Afzal MR, Gunda S, Waheed S, Sehar N, Maybrook RJ, Dawn B, Lakkireddy D. Role of Outpatient Cardiac Rhythm Monitoring in Cryptogenic Stroke: A Systematic Review and Meta-Analysis. Pacing Clin Electrophysiol. 2015 Oct;38(10):1236-45. doi: 10.1111/pace.12688. Epub 2015 Aug 27. PMID 26172621
- [Background] Ding EY, CastanedaAvila M, Tran KV, Mehawej J, Filippaios A, Paul T, Otabil EM, Noorishirazi K, Han D, Saczynski JS, Barton B, Mazor KM, Chon K, McManus DD. Usability of a smartwatch for atrial fibrillation detection in older adults after stroke. Cardiovasc Digit Health J. 2022 Apr 18;3(3):126-135. doi: 10.1016/j.cvdhj.2022.03.003. eCollection 2022 Jun. PMID 35720675
- [Background] Poli S, Diedler J, Hartig F, Gotz N, Bauer A, Sachse T, Muller K, Muller I, Stimpfle F, Duckheim M, Steeg M, Eick C, Schreieck J, Gawaz M, Ziemann U, Zuern CS. Insertable cardiac monitors after cryptogenic stroke--a risk factor based approach to enhance the detection rate for paroxysmal atrial fibrillation. Eur J Neurol. 2016 Feb;23(2):375-81. doi: 10.1111/ene.12843. Epub 2015 Oct 16. PMID 26470854